CLINICAL TRIAL: NCT02639533
Title: Pregabalin Acute Effects on Cortical Excitability, Psychophysical Parameters, and Serum Markers of Neuroplastic Processes in Fibromyalgia: a Placebo Controlled, Double Blinded, Randomized, Crossover Clinical Trial
Brief Title: Brain Response to Single Dose of Pregabalin in Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14-0624
Record Dates: First submitted 2015-11-11; First posted 2015-12-24 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2015-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pregabalin; cortical excitability; functional near infrared spectroscopy
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin 150 mg PO single dose
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Placebo (a pill of same physical characteristics as the one used for the experimental arm, containing starch) PO single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150 mg PO, single dose.
  Arms: Pregabalin
Other: Placebo — Pill of same physical characteristics as the one used for the intervention, containing starch only. Administered PO in single dose.
  Arms: Placebo

SUMMARY:
Fibromyalgia syndrome represents a "spectrum disorder" characterized by widespread chronic pain, fatigue, sleep disturbances, mood and cognitive alterations. The most accepted models explaining the causes of the disease have focused on the reduced pain inhibitory systems activity, that allow low intensity stimuli to be processed easier, and that finally amplify pain stimuli. One of the interventions approved for Fibromyalgia is Pregabalin, which demonstrated to be effective reducing pain. Different studies in animals have shown that it works reducing the liberation of neuronal messengers, which slow the conduction of pain signals. Although studies in humans have confirmed Pregabalin clinical benefits, there are still few studies aiming to explain how it actually works in patients with fibromyalgia, though.

A better understanding of the mechanisms by which Pregabalin reduces pain in patients with fibromyalgia would allow designing new interventions to enhance its clinical effects. Thus, the investigators propose to study in real-time the electrical, vascular and hormonal response of the brain of patients with fibromyalgia who receive a single dose of Pregabalin. The vascular response will be assessed using functional near infrared spectroscopy (fNIRS) neuroimaging techniques. The electrical response will be assessed using Transcranial Magnetic Stimulation (TMS). The hormonal response will be assessed in blood, measuring neurotrophins (Brain Derived Neurotrophic Factor) and inflammatory mediators (Tumor Necrosis Factor). These responses will be studied in consideration of the patients' characteristics that will be assessed using validated scales.

Taken into account the above considerations, a crossover, double-blinded randomized clinical trial is proposed. In the investigators' study, patients and healthy volunteers will be asked to visit the investigators' laboratory in three opportunities: one for a baseline assessment, and the other two to test the effects of either Pregabalin 150 mg PO or Placebo. All participants will eventually receive both, Pregabalin and Placebo. In each visit a brain hemodynamic, electrical, hormonal and clinical evaluation will be performed.

DETAILED DESCRIPTION:
A crossover, double-blinded randomized clinical trial is proposed. The investigators will recruit literate adult females aging 18 to 65 years old; fulfilling the diagnosis criteria for fibromyalgia according to the American College of Rheumatology 2010; with mean pain ≥6 in the verbal analog scale; who speak Brazilian Portuguese; and were able to perform the three visits. Female adult participants without chronic pain will also be recruited. Participants with severe psychiatric disorders that would limit consenting; neurologic deficits; decompensated systemic disease or chronic inflammatory disorders (Systemic Erythematous Lupus or Rheumatoid arthritis); contraindications for TMS; and those with previous use of Pregabalin will be excluded.

In the investigators' study, participants will be asked to visit the investigators' laboratory in three opportunities: one for a baseline assessment, and the other two to test the effects of either Pregabalin 150 mg PO or Placebo. All participants will eventually receive both, Pregabalin and Placebo. In each visit a brain hemodynamic, electrical, hormonal and clinical evaluation will be performed.

In the first visit, after explaining the research, solving doubts and signing the informed consent, participants will be randomized to an allocation sequence (either Pregabalin in the second or in the third visit). Then, a blood sample will be gathered and participants will be asked to fill some questionnaires to understand better their pain, and its impact on their quality of life (Fibromyalgia Impact Questionnaire), Anxiety (State/Trait Anxiety Inventory), Depressive symptoms (Beck Depression Inventory II), Catastrophizing thinking (Pain Catastrophizing Scale - PCS), Sleep (Pittsburgh Sleep Quality Index), and resiliency. Then, a fingertapping task will be performed while assessing hemodynamic changes using fNIRS. After that, heat perception will be tested using quantitative sensory testing (QST) and Conditioned Pain Modulation (CPM) with cold. Also, the pain pressure threshold (PPT) using a digital algometer will be evaluated. Finally, cortical excitability parameters (motor evoked potentials, intracortical facilitation and inhibition, and cortical silent period) will be determined using paired pulsed TMS.

In the second visit, according to the randomized allocation participants will receive either Pregabalin 150 mg PO or Placebo. Then, the M.I.N.I. International Neuropsychiatric Interview will be performed. One hour after taking the medication, the fNIRS, QST, CPM, PPT and TMS evaluations will be repeated, and a new blood sample will be collected. In the third visit, a blood sample will be gathered, followed by administration of the corresponding intervention according to the randomized allocation. Then, the pain level, PCS, STAI and International Physical Activity Questionnaire (IPAQ) will be asked again. One hour after taking the medication, the fNIRS, QST, CPM, PPT and TMS evaluations will be repeated, and a final blood sample will be collected. Participants' guess about blinding will be assessed after each intervention. All evaluators will remain blind to the allocation.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill ACR 2010 criteria for fibromyalgia diagnosis.
* Literate.
* Mean VAS for pain higher than 6 in the last 3 months.

Exclusion Criteria:

* Pregnancy or inadequate use of validated contraceptive method.
* Contraindications for Transcranial Magnetic Stimulation.
* Alcohol of drugs abuse in the last 6 months.
* Any severe neurological, neurosurgical, cardiac, endocrinological, or oncological disease (current or past).
* Decompensated chronic systemic disease.
* Previous use of Pregabalin.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cortical Excitability: Intracortical Inhibition. | 1 hour after intervention
  Cortical excitability parameters assessed non-invasively using paired-pulse Transcranial Magnetic Stimulation. Intracortical inhibition will be assessed using a conditioning stimuli of 80% of the motor threshold (MT) and a testing pulse of 120% the of the MT, with interstimuli interval (isi) of 2 and 4 microseconds. The Intracortical Inhibition corresponds to the ratio between the resultant potential and the motor evoked potential.
Cortical hemodynamics: Oxy-hemoglobin concentration (mM/L) | 1 hour after intervention
  Cortical hemodynamics assessed non-invasively using functional near infrared spectroscopy. Thanks to spectroscopy principles, it is possible to safety use a light beam in the infrared spectrum to infer the concentration of hemoglobin when bonded to oxygen. Its concentration is calculated in mM/L.

SECONDARY OUTCOMES:
Pain | 1 hour after intervention
  Assessed with the Visual Analog Scale
Heat Pain Threshold | 1 hour after intervention
  Assessed using quantitative sensory testing. Briefly, a thermode placed in subjects forearm is heated controlled by a computer. Subjects are instructed to report when perceiving the first pain. Temperatures in Celcius degrees are recorded.
Pressure Pain Threshold | 1 hour after intervention
  Assessed using a digital algometer. Briefly, progressive pressure is applied in subjects forearm until the first perception of pain is reported. The pressure of the first perception of pain are recorded in Kg/cm^2 .
Maximal Heat Pain Tolerance | 1 hour after intervention
  Assessed using quantitative sensory testing. Briefly, the thermode placed in subjects forearm is heated until subject reports maximum tolerated pain. A maximal temperature of 52 Celcius has been previously programmed for the device to stop and cool down in order to avoid unintended injuries.
Conditioned pain modulation | 1 hour after intervention
  The protocol for heat pain threshold is repeated while the contralateral hand is placed on iced water. The pain due to heat and cold reported on a Visual Analog Scale are recorded.
Serum Brain Derived Neurotrophic Factor (BDNF) | Baseline and 2 hours after intervention
  Blood samples will be gathered at baseline and 2 hours after receiving the intervention to quantify the serum BDNF concentration (ng/mL).
Serum Protein S100B | Baseline and 2 hours after intervention
  Blood samples will be gathered at baseline and 2 hours after receiving the intervention to quantify the serum S100B concentration (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD, PhD, Principal Investigator — HCPA

REFERENCES:
- [Derived] Deitos A, Soldatelli MD, Dussan-Sarria JA, Souza A, da Silva Torres IL, Fregni F, Caumo W. Novel Insights of Effects of Pregabalin on Neural Mechanisms of Intracortical Disinhibition in Physiopathology of Fibromyalgia: An Explanatory, Randomized, Double-Blind Crossover Study. Front Hum Neurosci. 2018 Nov 19;12:406. doi: 10.3389/fnhum.2018.00406. eCollection 2018. PMID 30510505